CLINICAL TRIAL: NCT06594523
Title: A Phase 3, Randomized, Double-blind, Placebo-controlled Study Evaluating the Safety and Efficacy of Denifanstat in Patients With Noncirrhotic Metabolic Dysfunction-associated Steatohepatitis (MASH) and F2/F3 Fibrosis (FASCINATE-3)
Brief Title: A Phase 3 Study Evaluating the Safety and Efficacy of Denifanstat in Patients With MASH and F2/F3 Fibrosis
Acronym: FASCINATE-3
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Business decision
Sponsor: Sagimet Biosciences Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SB2640-CLIN-010
Record Dates: First submitted 2024-09-10; First posted 2024-09-19 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: MASH; NASH; Metabolic Dysfunction-associated Steatohepatitis; Noncirrhotic Metabolic Dysfunction-associated Steatohepatitis; Nonalcoholic Steatohepatitis; Nonalcoholic Fatty Liver
Keywords: fibrosis; fatty liver; steatohepatitis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Fibrosis; Fatty Liver | interventions — TVB-2640

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Denifanstat 50 mg (Experimental): Denifanstat tablet, orally, once daily
  Interventions: Drug: Denifanstat
- Denifanstat 25 mg (Experimental): Denifanstat tablet, orally, once daily
  Interventions: Drug: Denifanstat
- Placebo (Placebo Comparator): Placebo tablet, orally, once daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Denifanstat — Tablet
  Other Names: TVB-2640
  Arms: Denifanstat 25 mg; Denifanstat 50 mg
Drug: Placebo — Matching Tablet
  Arms: Placebo

SUMMARY:
A randomized, double-blind, placebo-controlled Phase 3 study to determine if denifanstat 50 mg or 25 mg is effective, as compared to placebo, in resolving MASH without the worsening of fibrosis and/or in fibrosis regression without the worsening of steatohepatitis.

DETAILED DESCRIPTION:
Approximately 1260 patients (including at least 60% of F3 patients) will be enrolled to receive either denifanstat 50 mg (580 patients), placebo (580 patients), or denifanstat 25 mg (100 patients).

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to participate in the study and provide written informed consent.
2. Adults between 18 and 75 years of age.
3. Body mass index (BMI) ≥23 kg/m^2 for Asian patients and ≥25 kg/m^2 for patients of other races.
4. Presence of metabolic risk factor(s), as follows:

   1. T2DM.

      OR
   2. 2 out of 4 of the following:

      * BMI ≥30 kg/m^2.
      * Hypertension, or on active antihypertensive treatment.
      * Elevated fasting serum TGs or on active treatment for hypertriglyceridemia.
      * Reduced fasting serum HDL-c or on active treatment for dyslipidemia.
5. For patients with T2DM:

   * HbA1c ≤9.5%.
   * Metformin, insulin, dipeptidyl peptidase-4 inhibitors (DPP4-Is), sodium-glucose transport protein-2 inhibitors (SGLT2-Is), and alpha-glucosidase inhibitors (α-GIs): stable dose for at least 12 weeks prior to qualifying liver biopsy and screening.
   * Sulfonylureas (SUs) and glinides: stable dose with no history of relevant hypoglycemia for at least 12 weeks prior to qualifying liver biopsy and screening.
   * GLP-1 RA: stable dose for at least 18 weeks prior to start of screening.
6. Noncirrhotic, biopsy-proven MASH with:

   1. A fibrosis stage of F2 or F3.
   2. NAS ≥4 with at least a score of 1 in each of the following NAS components:

      * Steatosis (scored 0 to 3).
      * Hepatocyte ballooning (scored 0 to 2).
      * Lobular inflammation (scored 0 to 3).
7. A qualifying historical liver biopsy within 6 months before the screening visit. Historical biopsy results will be confirmed by central reading.

   If there is no available historical liver biopsy within this time period, a liver biopsy must be performed during the screening period. Patients should be deemed likely to have MASH F2/F3 fibrosis prior to proceeding to a liver biopsy, as indicated by the following:
   1. FibroScan.

      * Liver stiffness measurement (LSM) ≥8.5 kPa.
      * Controlled attenuation parameter (CAP) ≥280 dB/m.
   2. Aspartate aminotransferase (AST) >20 U/L.
8. Stable ALT and AST levels.

Exclusion Criteria:

1. Previous intake of an approved MASH medication.
2. Exclusionary laboratory values:

   1. ALT and/or AST >5 × ULN.
   2. ALP ≥2 × ULN.
   3. Total serum bilirubin concentration >1.3 mg/dL.
   4. Serum albumin concentration <3.5 g/dL.
   5. INR >1.3 except for patients receiving anticoagulant treatment.
   6. Platelet count <140,000/μL.
   7. Fasting TG level ≥500 mg/dL.
   8. eGFR <45 mL/min/1.73 m^2.
3. History of excessive alcohol intake for a period of more than 3 consecutive months within 1 year prior to screening.
4. Presence of cirrhosis on liver histology according to the assessment of the central reader.
5. Current or historical clinically evident hepatic decompensation.
6. Evidence of another form of active liver disease.
7. Positive serologic evidence of current infectious liver disease.
8. MELD score ≥12.
9. Planned or history of liver transplantation.
10. Prior or planned bariatric surgery.
11. Gain or loss of >5% of body weight in the 3 months or >10% of body weight in the 6 months prior to screening, qualifying liver biopsy, and the baseline visit (V1).
12. Any of the following within 6 months prior to the baseline visit (V1):

    1. Myocardial infarction.
    2. CABG/PTCA.
    3. Unstable angina.
    4. Transient ischemic attack, stroke, or cerebrovascular disease.
13. Unstable or undiagnosed arrhythmias.
14. Uncontrolled high BP.
15. Malignancy with a complete remission date within 5 years prior to the baseline visit (V1).
16. Any current or history of hepatocellular carcinoma.
17. Diabetes other than T2DM.
18. Uncontrolled hypothyroidism.
19. Any other known serious disease or other disease which in the Investigator's opinion would exclude the patient from participating in the study.
20. Previous intake of an approved MASH medication, unless there is at least a 6-month wash-out period between the last date of intake of the approved MASH medication and date of screening.
21. Use of a nonpermitted concomitant medication within 30 days or 5 half-lives prior to the qualifying liver biopsy and screening.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-03 (Estimated); Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Dual Primary Efficacy Endpoint 1: Interim Analysis: MASH Resolution (denifanstat 50 mg compared to placebo) | 52 weeks
  Proportion of patients who achieve MASH resolution (defined as NAS* of 0 for ballooning, and 0 or 1 for inflammation) without worsening of fibrosis stage at Week 52.
  *NAS: nonalcoholic fatty liver disease activity score
Dual Primary Efficacy Endpoint 2: Interim Analysis: Improvement in Fibrosis (denifanstat 50 mg compared to placebo) | 52 weeks
  Proportion of patients who achieve at least a 1-point improvement in fibrosis stage and without worsening of steatohepatitis (defined as no increase in NAS* for ballooning, inflammation, or steatosis) at Week 52.
Primary Endpoint: End of Study Analysis: Liver-related Composite Clinical Outcome (denifanstat 50 mg compared to placebo) | 234 weeks
  Time to first occurrence of any event from the following composite clinical outcome: death from any cause; histopathologic progression to cirrhosis; liver transplant; Model for End-Stage Liver Disease (MELD) score ≥15; Liver decompensation event defined by: Ascites requiring chronic diuretic treatment, Hepatic encephalopathy grade 2 or above requiring at least a 24-hour hospitalization, Variceal hemorrhage requiring hospitalization and transfusion of blood.

IPD SHARING:
Plan to Share IPD: No